CLINICAL TRIAL: NCT05552391
Title: Dexametomedine Versus Ketamine as an Adjuvant in Ultrasound Guided Erector Spinae Block for Perioperative Thoracotomy Pain Control in Pediatrics Cardiothoracic Surgeries: A Randomized Controlled Trial
Brief Title: Dexametomedine Versus Ketamine as an Adjuvant in Erector Spinae Block for Perioperative Thoracotomy Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Lecturer of Anesthesia, ICU and Pain managment, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-88-2022
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bupivacaine (Placebo Comparator): Group bupivacaine(Control) (B) received 0.5 ml/kg bupivacaine 0.25% diluted with isotonic saline (total volume15 ml).
  Interventions: Drug: Bupivacaine
- bupivacaine - ketamine (Active Comparator): Group bupivacaine - ketamine (K) received 0.5 ml/kg bupivacaine 0.25% with ketamine 2 mg/kg, diluted with isotonic saline (total volume15 ml).
  Interventions: Drug: Bupivacaine; Drug: Ketamine Hydrochloride
- bupivacaine - Dexametomedine (Active Comparator): Group bupivacaine - Dexametomedine (D) received 0.5 mL/kg bupivacaine 0.25% with dexmedetomidine 1 µg/kg. diluted with isotonic saline (total volume 15ml).
  Interventions: Drug: Bupivacaine; Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine — Group bupivacaine(Control) (B) received 0.5 ml/kg bupivacaine 0.25% diluted with isotonic saline (total volume15 ml).
  Other Names: Marcaine
Drug: Ketamine Hydrochloride — Group bupivacaine - ketamine (K) received 0.5 ml/kg bupivacaine 0.25% with ketamine 2 mg/kg, diluted with isotonic saline (total volume15 ml).
  Other Names: Ketalar
  Arms: bupivacaine - ketamine
Drug: Dexmedetomidine Hydrochloride — Group bupivacaine - Dexametomedine (D) received 0.5 mL/kg bupivacaine 0.25% with dexmedetomidine 1 µg/kg. diluted with isotonic saline (total volume 15ml).
  Other Names: Precedex
  Arms: bupivacaine - Dexametomedine

SUMMARY:
A double-blind randomized control study to compare the efficacy of dexmedetomidine versus ketamine as an adjuvant in combination with bupivacaine ultrasound-guided ESP block in patients scheduled for cardiothoracic surgeries with thoracotomy incision.

DETAILED DESCRIPTION:
Following approval from research and ethics committee ,preoperative preparation, and induction of anesthesia Patients will be allocated to three groups according to the type of drug injected.

Group bupivacaine(Control) (B) received 0.5 ml/kg bupivacaine 0.25% diluted with isotonic saline (total volume15 ml).

Group bupivacaine - ketamine (K) received 0.5 ml/kg bupivacaine 0.25% with ketamine 2 mg/kg, diluted with isotonic saline (total volume15 ml).

Group bupivacaine - Dexametomedine (D) received 0.5 mL/kg bupivacaine 0.25% with dexmedetomidine 1 µg/kg. diluted with isotonic saline (total volume 15ml).

Unilateral Ultrasound-guided erector spinae block will be applied in both groups after the induction of anaesthesia. All patients will be tilted onto their left side (lateral position). while the ultrasound-guide unilateral erector spinae block will be performed under completely aseptic conditions. The anatomy will be examined by ultrasonography at 5-6Hz with a35 mm linear probe and a SonoSite M-turbo system (Fujifilm SonoSite, Inc., USA). a 22 g bevel needle will be advanced in a cephalad to caudad direction until the tip of the needle reach' the plane deep to the erector spinae muscle and immediately lateral to the transverse process. Once confirmed, after careful aspiration to demonstrate the absence of air or blood. An injection in this plane permitted the block to impact both the dorsal and ventral rami as they exited from the thoracic spine to innervate the chest wall. the block permits a diminished sensation spanning the T3-T10 dermatome levels. confirming the correct tissue plane by hydro-dissection.

Heart rate, mean arterial pressure, and oxygen saturation will be monitored continuously.

After completion of the surgery, inhalational anesthetics will be stopped as well the muscle relaxant. The patient will be then transferred to the ICU.

Postoperative assessment and analgesic regimen:

Post-operative pain intensity will be assessed using the objective pain score (OPS) by a person who will be blinded to the treatment. OPS score will be recorded at baseline,3,6,12,24 and 48 hours post-operatively to evaluate acute pain will be observed and recorded. for the score 4 or more, which was considered the end point of the study, and at this point. Patients will receiv paracetamol 15 gm / Kg IV /6 h, as components of multimodal analgesia regimen for postoperative pain control.

Persistent or breakthrough pain will be managed with incremental intravenous morphine at a dose of 0.1mg/kg to maintain resting (OPS) score ˂ 4.

ELIGIBILITY:
Inclusion Criteria:

* age from 3 to 36 months
* weight >5 kg.
* gender both males and females
* cardiothoracic surgeries with thoracotomy incision.

Exclusion Criteria:

* 1 Skin erosions , hematomas or infection at or near the injection site.
* 2. coagulopathy,
* 3. History of hypersensitivity to bupivacaine ,ketamine or dexametomedine.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
the duration of analgesia | immediately at the end of pediatric cardiac operation
  the duration of analgesia from block start time (time of LA injection) to block end time at which OPS score 4 or more) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided